CLINICAL TRIAL: NCT03474978
Title: Peripherally Inserted Central Venous Catheter Insertion Site and Complication Rates in Neonates
Brief Title: Peripherally Inserted Central Catheter Insertion Site and Complication Rate in Neonates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Amuchou Soraisham, Neonatologist, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB17-2371
Record Dates: First submitted 2018-03-14; First posted 2018-03-23 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Catheterization, Peripheral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Upper Extremity Insertion (Experimental): Peripherally Inserted Central Venous Cather (PICC) inserted in upper extremity
  Interventions: Device: Peripherally Inserted Central Venous Cather (PICC)
- Lower Extremity Insertion (Experimental): Peripherally Inserted Central Venous Cather (PICC) inserted in lower extremity
  Interventions: Device: Peripherally Inserted Central Venous Cather (PICC)

INTERVENTIONS:
Device: Peripherally Inserted Central Venous Cather (PICC) — Location of the PICC insertion will be randomized and compared

SUMMARY:
This study examines whether there is an association between the PICC insertion site and the complications necessitating PICC removal in neonates admitted to neonatal intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

1. Neonates of all gestational ages admitted to Foothills Medical Centre and Alberta Children's Hospital Neonatal Intensive Care Unit (NICU)
2. Peripherally inserted central venous catheter (PICC) line insertion planned as part of NICU care
3. Venous access available in both upper(above umbilicus) and lower body

Exclusion Criteria:

1. Local infection at potential site of insertion
2. Hemangioma, lymphangioma or malformations in the region of insertion
3. Major chromosomal anomalies

Max Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 320 (Estimated)
Dates: Start 2018-10-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary outcome is the presence of any complication which necessitates PICC removal | Through study completion, within 4 weeks
  Line infiltration will be defined as extravasation of fluid into soft tissue around the region of the catheter tip. Line occlusion will be defined as inability to infuse fluid, resulting in removal of line. Phlebitis will be defined as presence of a linear red streak developing along the superficial veins from the catheter insertion site. Line associated thrombosis will be defined as ultrasound proven evidence of an occlusive thrombus in an anatomic location in proximity to the site of PICC.CLABSI will be defined according to Center for Disease Control definitions 26, that is, (1) confirmed primary bloodstream infection with (2) one of following clinical signs of infection (fever, hypothermia, apnea, or bradycardia) and (3) presence of central catheter at the time of or within 48 hours before the onset of the infection. Major life-threatening complications will include pleural effusion, pericardial effusion and cardiac tamponade, retroperitoneal extravasation.

SECONDARY OUTCOMES:
Secondary outcome will be time to complication post insertion | Through study completion, within 4 weeks
  This will be defined as the interval between PICC line insertion and first detection of complication post insertion, expressed in days.

CONTACTS AND LOCATIONS:
Overall Officials: Amuchou Soraisham, MD, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-12-05): https://cdn.clinicaltrials.gov/large-docs/78/NCT03474978/Prot_SAP_000.pdf
  • Informed Consent Form (2018-03-02): https://cdn.clinicaltrials.gov/large-docs/78/NCT03474978/ICF_001.pdf